CLINICAL TRIAL: NCT05748327
Title: Randomized Controlled Clinical Trial (RCT) of the New Tooth-colored Restorative Material 'Cention Forte' (Ivoclar Vivadent) vs. 'Equia Forte HT' (GC) in Class-I/II Cavities
Brief Title: Trial With Two New Tooth-colored Restorative Materials in Class I/II Cavities
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ivoclar Vivadent AG (Industry)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LL4199644; S66086 (Other: KU Leuven)
Record Dates: First submitted 2023-02-09; First posted 2023-02-28 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Caries; Defective Restorations

STUDY DESIGN:
Intervention Model Description: Split-Mouth Design
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Alcasite restorative material (Experimental)
  Interventions: Device: Alcasite restorative material
- Bulk fill glass hybrid restorative material (Active Comparator)
  Interventions: Device: Bulk fill glass hybrid restorative material

INTERVENTIONS:
Device: Alcasite restorative material — Cavity preparation, pulp protection (if necessary), placing matrix/ interdental wedge (if necessary), conditioning with primer, mixing alcasite capsula, place restoration, polymerizing and finishing
  Arms: Alcasite restorative material
Device: Bulk fill glass hybrid restorative material — Cavity preparation, pulp protection (if necessary), placing matrix/ interdental wedge (if necessary), mixing bulk fill glass hybrid capsula, conditioning, place restoration, apply coating, polymerizing and finishing
  Arms: Bulk fill glass hybrid restorative material

SUMMARY:
This is a randomized-controlled clinical trial to investigate the success rate of two new tooth-colored restorative materials in class I and II cavities over 5 years according to FDI criteria scores (1, 2 and 3).

DETAILED DESCRIPTION:
The primary outcome of the study is the SUCCESS RATE of restorations placed with both filling materials in class I and II cavities after 5 years of clinical service. A failure which leads to repair or replacement of the restoration can have esthetic (marginal staining, loss of anatomical form), functional (i.e. fracture of restoration, loss of retention) or biological reasons (i.e. secondary caries). A restoration is defined as a failure (no success) as soon as at least one FDI criterion is scored as 4 or 5.

ELIGIBILITY:
Inclusion Criteria:

* Subject's age between 18 and 65 years old
* Class I and Class II (with a cavity margin 1-1.5 mm from the cusp tip) (caries treatment, removal of existing defective amalgam/composite restorations), on premolars/molars
* Vital teeth
* 2 restorations per patient: both cavities should have comparable size and dimensions
* Presence of neighbour tooth and antagonist (molars with no neighbour tooth at the distal side can also be included)
* Low to moderate caries rate/normal periodontal status with good home care

Exclusion Criteria:

* Hospitalized and medically compromised patients (medical history may not compromise the outcome of the results)
* Pulp exposure or signs of pulpal infection
* No signs of pulpitis or hypersensitivity (Visual analog scale < 3 on biting and temperature sensitivity)
* History of allergy to glass ionomer, acrylate/methacrylate monomers
* Pregnancy
* Chronic disease with oral manifestations or primary oral pathology
* Bad oral hygiene
* High caries rate or periodontal problems
* Absence of antagonists
* Absence of adjacent teeth (except last molar in the row with no neighbour tooth at the distal side)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2022-11-22 (Actual); Primary Completion 2028-04-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Success Rate | 5 years
  assessed following FDI criteria on a scale from 1 "very good" to 5 "unacceptable": e.g. post-operative hypersensitivity, surface lustre, staining, fracture of material, retention, occlusal contour and wear, and colour match of restorations (Success: Scores equal to/above 3)

SECONDARY OUTCOMES:
Success Rate | 6 months to 3 years
  assessed following FDI criteria on a scale from 1 "very good" to 5 "unacceptable": e.g. post-operative hypersensitivity, surface lustre, staining, fracture of material, retention, occlusal contour and wear, and colour match of restorations (Success: Scores equal to/above 3)
Survival Rate | 6 months to 5 years
  assessed following FDI criteria on a scale from 1 "very good" to 5 "unacceptable": e.g. post-operative hypersensitivity, surface lustre, staining, fracture of material, retention, occlusal contour and wear, and colour match of restorations (Survival: Score equal to/above 4)
Quality criteria (Clinical performance) | 6 months to 5 years
  assessed following FDI criteria on a scale from 1 "very good" to 5 "unacceptable": e.g. post-operative hypersensitivity, surface lustre, staining, fracture of material, retention, occlusal contour and wear, and colour match of restorations

CONTACTS AND LOCATIONS:
Locations (1):
- KU Leuven, Leuven, Belgium